CLINICAL TRIAL: NCT06929806
Title: A Phase III, Randomized, Open-label, Blinded Endpoint, Comparative Trial of Ferric Derisomaltose Versus no Intravenous Iron in Iron-deficient Subjects With Symptomatic Chronic Heart Failure
Brief Title: Multi-center Trial of Ferric Derisomaltose Versus no Intravenous Iron in Iron-deficient Subjects With Symptomatic Chronic Heart Failure
Acronym: ICONIC-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-Monofer-CHF-02
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Chronic Heart Failure; Iron Deficiencies
MeSH Terms: conditions — Iron Deficiencies | interventions — ferric derisomaltose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferric Derisomaltose (Experimental): 50 % of the subjects will be treated with Ferric Derisomaltose 100 mg/mL The ferric derisomaltose dose administered is dependent on the subject's weight and hemoglobin (Hb) level. Subjects treated with ferric derisomaltose will be eligible for re-dosing if transferrin saturation (TSAT) remains below <25 %
  Interventions: Drug: Ferric Derisomaltose
- Control (No Intervention): 50 % of the subjects will receive no IV iron

INTERVENTIONS:
Drug: Ferric Derisomaltose — 100 mg/mL
  Arms: Ferric Derisomaltose

SUMMARY:
The goal of this clinical trial is to learn if the IV Iron treatment ferric derisomaltose helps in the treatment of chronic heart failure in people with iron deficiency. The main question it aims to answer is:

• How many participants are admitted to the hospital or die from a disease in the heart or blood vessels

Researchers will compare treatment with ferric derisomaltose to no treatment with ferric derisomaltose. This will be done to see how well ferric derisomaltose works.

Participants will:

* Be randomized 50/50 to either treatment with Ferric derisomaltose or to no treatment with ferric derisomaltose
* All participants receives standard of care
* Visit site 4-5 times and have 7 video/phone-calls

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Both women and men can join
* Heart failure that causes fatigue, shortness of breath, or other symptoms during physical activity
* Have left ventricle (chamber) ejection fraction (pumping ability) that is 45% or less
* Have low iron levels in the blood
* New York Heart Association (NYHA) Heart Failure Classification II, III or IV

Exclusion Criteria:

* Planned cardiac surgery or revascularization or cardiac device implantation
* Pregnant or nursing women
* Treatment with iron Intravenous (through the vein) or intramuscular (injection in the muscle) within the past 6 months
* Treatment with radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular deaths and hospitalizations for worsening heart failure | From enrollment to the end of follow-up at 52 weeks

SECONDARY OUTCOMES:
Number of hospitalizations for worsening heart failure | From enrollment and no longer than end of follow-up at 52 weeks
Time to cardiovascular death | From enrollment to the end of follow-up at 52 weeks
Number of all-cause hospitalizations | From enrollment to the end of follow-up at 52 weeks
Time to all-cause death | From enrollment to the end of follow-up at 52 weeks
Time to first hospitalization for worsening heart failure or cardiovascular death | From enrollment to the end of follow-up at 52 weeks
Number of hospitalizations for cardiovascular, respiratory, or renal disease | From enrollment to the end of follow-up at 52 weeks
Time to cardiovascular, respiratory, or renal death | From enrollment to the end of follow-up at 52 weeks
Number of hospitalizations for cardiovascular events: stroke, AMI and heart failure | From enrollment to the end of follow-up at 52 weeks
Time to cardiovascular death or first hospitalization for cardiovascular event: stroke, AMI and heart failure | From enrollment to the end of follow-up at 52 weeks
Time to all-cause death or first hospitalization | From enrollment to the end of follow-up at 52 weeks
Days hospitalized or dead for cardiovascular reasons at week 52 | From enrollment to the end of follow-up at 52 weeks
Days hospitalized or dead for any reason at week 52 | From enrollment to the end of follow-up at 52 weeks
Change in NYHA from baseline to weeks 12, 26 and 52 | From enrollment to weeks 12, 26 and 52
All-cause rehospitalizations at 30 and 60 days | From enrollment to 30 and 60 days
Rehospitalizations for worsening heart failure at 30 and 60 days | From enrollment to 30 and 60 days
Number of cardiovascular deaths and hospitalizations for worsening heart failure including urgent and unscheduled outpatient IV diuretic treatment | From enrollment to the end of follow-up at 52 weeks
Number of urgent and unscheduled outpatient IV diuretic treatment | From enrollment to the end of follow-up at 52 weeks

OTHER OUTCOMES:
Change in hb, s-ferritin, TSAT, s-iron and TIBC from baseline to weeks 26 and 52 | From enrollment to weeks 26 and 52
Type and incidence of SAEs | From enrollment to the end of follow-up at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos Clinical and non-clinical department, Study Director — Pharmacosmos A/S
Locations (1):
- Private clinic, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No